CLINICAL TRIAL: NCT06350578
Title: Comparative Analysis of Hall Technique and Conventional Method for Stainless Steel Crown Placement in Primary Molars With Approximal Caries: A Randomized Controlled Trial at Primary Healthcare Corporation, Qatar
Brief Title: A Randomized Clinical Trial Comparing Hall vs. Conventional Technique in Primary Molars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primary Health Care Corporation, Qatar (Other Government)
Responsible Party: Principal Investigator, Hanan Mohamed, Pediatric Dentistry Specialist, Primary Health Care Corporation, Qatar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUHOOTH-D-23-00073
Record Dates: First submitted 2024-03-24; First posted 2024-04-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-03

CONDITIONS: Approximal Dental Caries (ICDAS 3-5) in Primary Molars of Children
Keywords: Hall Technique; Conventional Restoration; Stainless Steel Crowns; Approximal Caries; Paediatric Dentistry; Non-inferiority Trial; Minimally Invasive Dentistry; Pain Perception; Parental Acceptability; Occlusal Vertical Dimension; Restoration Survival; Tooth Survival; Randomised Controlled Trial

STUDY DESIGN:
Intervention Model Description: A binary outcome non-inferiority randomised trial.
Who Masked: Care Provider
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hall Crown Technique (Experimental): HT is a conservative restorative technique used for primary molars with single- or multi-surface carious lesions. This technique involves cementing a SSC directly over the affected primary molar without any caries removal or tooth reduction.
  Interventions: Procedure: Hall Crown Technique
- Conventional SSC Technique (Active Comparator): CT is the traditional restorative technique often used for primary molars with multi-surface carious lesions. This technique involves caries removal and occlusal-proximal tooth surface reduction before crown cementation.
  Interventions: Procedure: Conventional SSC Technique

INTERVENTIONS:
Procedure: Hall Crown Technique — The Hall technique (HT) involves cementing Stainless Steel Crowns SSC on carious primary teeth without using rotary instruments nor local anaesthesia, thus eliminating discomfort, and increasing child's behavior.
  Arms: Hall Crown Technique
Procedure: Conventional SSC Technique — The conventional technique involves complete removal of the carious lesion using rotary instruments and local anesthesia, then restoring the tooth with Stainless Steel Crown SSC.
  Arms: Conventional SSC Technique

SUMMARY:
This study aims to assess the comparative effectiveness of the Hall technique (HT) and the conventional technique (CT) for placing Stainless Steel Crowns (SSCs) in primary molars with approximal caries.

DETAILED DESCRIPTION:
Background:

The most common chronic disease in children and adolescents (6-19 years old) is dental caries. The conventional approach to treating carious lesions involves cavity preparation with rotary instruments, followed by restoration using composite resin, amalgam, or stainless steel crowns (SSCs).

Retrospective studies have shown that SSCs have a higher success rate compared to amalgam or resin-based restorations when used for multi-surface caries in primary teeth. Accordingly, the American Academy of Paediatric Dentistry (AAPD) recommends the use of SSCs as the treatment of choice for carious lesions involving more than one surface in high-risk children.

Recently, the Hall Technique (HT) has been used to seal caries in primary molars. This contemporary technique was first introduced in the literature in 2006 by Dr Norna Hall, while working in a high caries-risk area in rural Scotland. The technique is based on straightforward biological principles: the most important layer for caries progression- the superficial plaque layer- is left intact and sealed along with the carious lesion. This leads to the development of a less cariogenic flora within the plaque biofilm, thereby arresting or slowing the caries progression in primary teeth.

The Hall Technique involves cementing an SSC over a carious primary tooth without the use of rotary instruments or local anaesthesia, thus reducing discomfort and improving the child's behaviour during treatment.

Aim:

The study aims to compare the Hall Technique (HT) and Conventional Restoration (CR) using stainless steel crowns (SSCs) in terms of clinical effectiveness, changes in occlusal vertical dimension (OVD), procedural time, child pain perception and cooperation, as well as parental acceptability of both techniques.

Methods/Design:

Approximal dental caries (ICDAS 3-5) in primary molars of children aged 3 to 9 years will be managed using two treatment techniques: conventional restorations (CR) with stainless steel crowns (SSCs) and the Hall Technique (HT). The study will be a binary outcome, non-inferiority randomised trial conducted in a primary care dental clinic setting. The study protocol will follow the Consolidated Standards of Reporting Trials (CONSORT) guidelines for randomised trials of non-pharmacologic treatments. Participants will be randomly allocated to receive SSCs placed using either the conventional technique (CT, control group) or the Hall Technique (HT, experimental group), in order to compare different approaches for managing occluso-proximal caries lesions in primary molars.

Discussion:

This clinical trial aims to determine whether the Hall Technique (HT) provides clinical outcomes that are not inferior to those of conventional restorations (CR) using stainless steel crowns (SSCs) in the management of approximal caries in primary molars. The study will also assess child pain perception, cooperation, and parental acceptability, to support the use of minimally invasive techniques in paediatric dental care.

ELIGIBILITY:
Inclusion Criteria:

* Participant inclusion criteria:

PHCC paediatric dental patients:

1. Whose parents or legal guardians accept and sign the consent form
2. Who assent to participation.
3. Who aged 3-9 years old.
4. Who exhibit generally cooperative behavior.
5. Who exhibit good general health conditions.
6. Who are presenting at least one occluso-proximal lesion in a primary molar.

Tooth/ carious lesion inclusion criteria:

1. From clinical and radiographic examination, caries limited to the occluso-proximal surfaces and extending to enamel or dentine, cavitated or non cavitated.

Exclusion Criteria:

1. Uncooperative children who do not understand the procedure or tolerate biting the crown into its position without local anesthesia.
2. Children with special health care needs (SHCN) will be excluded.
3. Children with nickel allergies and sensitivity.

Tooth/ caries lesion exclusion criteria:

1. Tooth with signs or symptoms of dental infection or irreversible pulpitis such as:

   A history of spontaneous unprovoked pain, a sinus tract, soft tissue inflammation not resulting from gingivitis or periodontitis, excessive mobility not associated with trauma or exfoliation, furcation/ apical radiolucency, or radiographic evidence of internal/ external resorption (Camp JH 2011).
2. Crowns severely destructed with caries, which considered non-restorable (Innes, N.P 2009).
3. Teeth with single surface (occlusal) caries.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Restoration survival over 12 months | At 1 month, 6 months, 9 months, and 12 months post-treatment
  Success:
  * Satisfactory restoration/crown, no intervention required
  * No clinical or radiographic signs or symptoms of pulp pathology
  * Tooth exfoliated
  Minor Failures:
  * Secondary caries or new lesions detected clinically
  * Crown presents perforation
  * Restoration fracture or wear - intervention required
  * Loss of restoration - tooth that can be re-restored
  * Crown loss - tooth able to be re-treated
  * Reversible pulpitis, which could be treated without the need for extraction or pulpotomy
  Major Failures:
  * Irreversible pulpitis or dental fistula/abscess requiring pulpotomy or extraction
  * Loss of restoration/crown - tooth not capable of being re-restored
  * Periradicular and/or furcation radiolucency
Occlusal Vertical Dimension (OVD) resolution | Assessments will be conducted at baseline (before treatment), immediately after crown placement, and at follow-up visits at 1, 6, 9, and 12 months post-treatment, with particular emphasis on the 1-month follow-up.
  Will be assessed only in the HT group using a millimetre dental probe.

SECONDARY OUTCOMES:
Tooth survival over 12 months | At 1 month, 6 months, 9 months, and 12 months post-treatment
  Teeth with treatments scored as satisfactory or with minor failures will be classified as "successful," while teeth presenting major failures will be considered as "failure for tooth." Data related to the treated tooth will be collected for both groups.
Procedural Time | At the time of treatment visit
  Will be recorded during the treatment visit using a stopwatch for both the Hall Technique and the Conventional Technique.
Participant's cooperation | At the time of treatment visit
  Participant cooperation will be assessed and compared between the two intervention groups using the Frankl Behaviour Rating Scale.
Participant's pain perception | At the time of treatment visit
  Pain perception will be assessed and compared between the two intervention groups using the Wong-Baker Faces Pain Scale (WBFPS).
Parents' perceptions and opinions regarding treatment | At the time of treatment visit
  A five-point Likert scale will be used to assess the following:
  * Child's behaviour during treatment
  * Comfort during treatment
  * Satisfaction with treatment undertaken
  * Dentist's ease of treatment provision
  * Perceived duration of the procedure
  * Willingness to choose the same treatment option again

CONTACTS AND LOCATIONS:
Overall Officials: Hanan A Mohamed, Principal Investigator — Primary Health Care Corporation (PHCC) of Qatar
Locations (1):
- Primary Healthcare Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alshoraim MA, El-Housseiny AA, Farsi NM, Felemban OM, Alamoudi NM, Alandejani AA. Effects of child characteristics and dental history on dental fear: cross-sectional study. BMC Oral Health. 2018 Mar 7;18(1):33. doi: 10.1186/s12903-018-0496-4. PMID 29514657
- [Background] Araujo MP, Innes NP, Bonifacio CC, Hesse D, Olegario IC, Mendes FM, Raggio DP. Atraumatic restorative treatment compared to the Hall Technique for occluso-proximal carious lesions in primary molars; 36-month follow-up of a randomised control trial in a school setting. BMC Oral Health. 2020 Nov 11;20(1):318. doi: 10.1186/s12903-020-01298-x. PMID 33176756
- [Background] Ayedun OS, Oredugba FA, Sote EO. Comparison of the treatment outcomes of the conventional stainless steel crown restorations and the hall technique in the treatment of carious primary molars. Niger J Clin Pract. 2021 Apr;24(4):584-594. doi: 10.4103/njcp.njcp_460_20. PMID 33851682
- [Background] Badar SB, Tabassum S, Khan FR, Ghafoor R. Effectiveness of Hall Technique for Primary Carious Molars: A Systematic Review and Meta-analysis. Int J Clin Pediatr Dent. 2019 Sep-Oct;12(5):445-452. doi: 10.5005/jp-journals-10005-1666. PMID 32440052
- [Background] Barretto Ede P, Ferreira e Ferreira E, Pordeus IA. Evaluation of toothache severity in children using a visual analogue scale of faces. Pediatr Dent. 2004 Nov-Dec;26(6):485-91. PMID 15646909
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Methods and processes of the CONSORT Group: example of an extension for trials assessing nonpharmacologic treatments. Ann Intern Med. 2008 Feb 19;148(4):W60-6. doi: 10.7326/0003-4819-148-4-200802190-00008-w1. PMID 18283201
- [Background] Boyd DH, Page LF, Thomson WM. The Hall Technique and conventional restorative treatment in New Zealand children's primary oral health care - clinical outcomes at two years. Int J Paediatr Dent. 2018 Mar;28(2):180-188. doi: 10.1111/ipd.12324. Epub 2017 Aug 8. PMID 28787534
- [Background] Boyd DH, Thomson WM, Leon de la Barra S, Fuge KN, van den Heever R, Butler BM, Leov F, Foster Page LA. A Primary Care Randomized Controlled Trial of Hall and Conventional Restorative Techniques. JDR Clin Trans Res. 2021 Apr;6(2):205-212. doi: 10.1177/2380084420933154. Epub 2020 Jun 19. PMID 32559403
- [Background] Chua DR, Tan BL, Nazzal H, Srinivasan N, Duggal MS, Tong HJ. Outcomes of preformed metal crowns placed with the conventional and Hall techniques: A systematic review and meta-analysis. Int J Paediatr Dent. 2023 Mar;33(2):141-157. doi: 10.1111/ipd.13029. Epub 2022 Oct 17. PMID 36151937
- [Background] Ebrahimi M, Shirazi AS, Afshari E. Success and Behavior During Atraumatic Restorative Treatment, the Hall Technique, and the Stainless Steel Crown Technique for Primary Molar Teeth. Pediatr Dent. 2020 May 15;42(3):187-192. PMID 32522320
- [Background] Elamin F, Abdelazeem N, Salah I, Mirghani Y, Wong F. A randomized clinical trial comparing Hall vs conventional technique in placing preformed metal crowns from Sudan. PLoS One. 2019 Jun 3;14(6):e0217740. doi: 10.1371/journal.pone.0217740. eCollection 2019. PMID 31158253
- [Background] Erdemci ZY, Cehreli SB, Tirali RE. Hall versus conventional stainless steel crown techniques: in vitro investigation of marginal fit and microleakage using three different luting agents. Pediatr Dent. 2014 Jul-Aug;36(4):286-90. PMID 25197992
- [Background] Eriksson AL, Paunio P, Isotupa K. Restoration of deciduous molars with ion-crowns: retention and subsequent treatment. Proc Finn Dent Soc. 1988;84(2):95-9. No abstract available. PMID 3134654
- [Background] Fayle SA. UK National Clinical Guidelines in Paediatric Dentistry. Stainless steel preformed crowns for primary molars. Faculty of Dental Surgery, Royal College of Surgeons. Int J Paediatr Dent. 1999 Dec;9(4):311-4. doi: 10.1046/j.1365-263x.1999.00153.x. No abstract available. PMID 10815591
- [Background] Frencken JE. Atraumatic restorative treatment and minimal intervention dentistry. Br Dent J. 2017 Aug 11;223(3):183-189. doi: 10.1038/sj.bdj.2017.664. PMID 28798450
- [Background] Frencken JE, Peters MC, Manton DJ, Leal SC, Gordan VV, Eden E. Minimal intervention dentistry for managing dental caries - a review: report of a FDI task group. Int Dent J. 2012 Oct;62(5):223-43. doi: 10.1111/idj.12007. PMID 23106836
- [Background] Hesse D, de Araujo MP, Olegario IC, Innes N, Raggio DP, Bonifacio CC. Atraumatic Restorative Treatment compared to the Hall Technique for occluso-proximal cavities in primary molars: study protocol for a randomized controlled trial. Trials. 2016 Mar 31;17:169. doi: 10.1186/s13063-016-1270-z. PMID 27029801
- [Background] Hu S, BaniHani A, Nevitt S, Maden M, Santamaria RM, Albadri S. Hall technique for primary teeth: A systematic review and meta-analysis. Jpn Dent Sci Rev. 2022 Nov;58:286-297. doi: 10.1016/j.jdsr.2022.09.003. Epub 2022 Sep 27. PMID 36185501
- [Background] Hussein I, Al Halabi M, Kowash M, Salami A, Ouatik N, Yang YM, Duggal M, Chandwani N, Nazzal H, Albadri S, Roberts A, Al-Jundi S, Nzomiwu C, El Shahawy O, Attaie A, Mohammed O, Al-Sane M. Use of the Hall technique by specialist paediatric dentists: a global perspective. Br Dent J. 2020 Jan;228(1):33-38. doi: 10.1038/s41415-019-1100-2. PMID 31925371
- [Background] Innes NP, Evans DJ, Stirrups DR. Sealing caries in primary molars: randomized control trial, 5-year results. J Dent Res. 2011 Dec;90(12):1405-10. doi: 10.1177/0022034511422064. Epub 2011 Sep 15. PMID 21921249
- [Background] Innes NP, Stirrups DR, Evans DJ, Hall N, Leggate M. A novel technique using preformed metal crowns for managing carious primary molars in general practice - a retrospective analysis. Br Dent J. 2006 Apr 22;200(8):451-4; discussion 444. doi: 10.1038/sj.bdj.4813466. PMID 16703041
- [Background] Innes NP, Evans DJ, Stirrups DR. The Hall Technique; a randomized controlled clinical trial of a novel method of managing carious primary molars in general dental practice: acceptability of the technique and outcomes at 23 months. BMC Oral Health. 2007 Dec 20;7:18. doi: 10.1186/1472-6831-7-18. PMID 18096042
- [Background] Kidd EA. How 'clean' must a cavity be before restoration? Caries Res. 2004 May-Jun;38(3):305-13. doi: 10.1159/000077770. PMID 15153704
- [Background] Kindelan SA, Day P, Nichol R, Willmott N, Fayle SA; British Society of Paediatric Dentistry. UK National Clinical Guidelines in Paediatric Dentistry: stainless steel preformed crowns for primary molars. Int J Paediatr Dent. 2008 Nov;18 Suppl 1:20-8. doi: 10.1111/j.1365-263X.2008.00935.x. PMID 18808544
- [Background] Ludwig KH, Fontana M, Vinson LA, Platt JA, Dean JA. The success of stainless steel crowns placed with the Hall technique: a retrospective study. J Am Dent Assoc. 2014 Dec;145(12):1248-53. doi: 10.14219/jada.2014.89. PMID 25429038
- [Background] Makansi N, Carnevale FA, Macdonald ME. The conceptualization of childhood in North American pediatric dentistry texts: a discursive case study analysis. Int J Paediatr Dent. 2018 Mar;28(2):189-197. doi: 10.1111/ipd.12325. Epub 2017 Aug 25. PMID 28840947
- [Background] Midani R, Splieth CH, Mustafa Ali M, Schmoeckel J, Mourad SM, Santamaria RM. Success rates of preformed metal crowns placed with the modified and standard hall technique in a paediatric dentistry setting. Int J Paediatr Dent. 2019 Sep;29(5):550-556. doi: 10.1111/ipd.12495. Epub 2019 Apr 14. PMID 30888708
- [Background] Nainar SM. Success of Hall technique crowns questioned. Pediatr Dent. 2012 Mar-Apr;34(2):103. PMID 22583879
- [Background] Roberts A, McKay A, Albadri S. The use of Hall technique preformed metal crowns by specialist paediatric dentists in the UK. Br Dent J. 2018 Jan 12;224(1):48-52. doi: 10.1038/sj.bdj.2018.4. PMID 29326453
- [Background] Rosenblatt A. The Hall technique is an effective treatment option for carious primary molar teeth. Evid Based Dent. 2008;9(2):44-5. doi: 10.1038/sj.ebd.6400579. PMID 18584001
- [Background] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Alkilzy M, Splieth CH. Acceptability of different caries management methods for primary molars in a RCT. Int J Paediatr Dent. 2015 Jan;25(1):9-17. doi: 10.1111/ipd.12097. Epub 2014 Mar 7. PMID 24602167
- [Background] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Splieth CH. Caries management strategies for primary molars: 1-yr randomized control trial results. J Dent Res. 2014 Nov;93(11):1062-9. doi: 10.1177/0022034514550717. Epub 2014 Sep 12. PMID 25216660
- [Background] Schwendicke F, Krois J, Robertson M, Splieth C, Santamaria R, Innes N. Cost-effectiveness of the Hall Technique in a Randomized Trial. J Dent Res. 2019 Jan;98(1):61-67. doi: 10.1177/0022034518799742. Epub 2018 Sep 14. PMID 30216734
- [Background] Schwendicke F, Stolpe M, Innes N. Conventional treatment, Hall Technique or immediate pulpotomy for carious primary molars: a cost-effectiveness analysis. Int Endod J. 2016 Sep;49(9):817-826. doi: 10.1111/iej.12537. Epub 2015 Sep 19. PMID 26331379
- [Background] van Amerongen WE, Rahimtoola S. Is ART really atraumatic? Community Dent Oral Epidemiol. 1999 Dec;27(6):431-5. doi: 10.1111/j.1600-0528.1999.tb02044.x. PMID 10600077
- [Background] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- See also: Behavior Guidance for the Pediatric Dental Patient — https://www.aapd.org/research/oral-health-policies--recommendations/behavior-guidance-for-the-pediatric-dental-patient/
- See also: Paediatric Restorative Dentistry — https://www.aapd.org/research/oral-health-policies--recommendations/pediatric-restorative-dentistry/
- See also: HALL TECHNIQUE VERSUS THE CONVENTIONAL STAINLESS STEEL CROWNS RESTORING CARIOUS PRIMARY MOLAR TEETH: A RANDOMIZED CONTROLLED CLINICAL TRIAL — https://www.semanticscholar.org/paper/HALL-TECHNIQUE-VERSUS-THE-CONVENTIONAL-STAINLESS-A-Sharaf-Dowidar/57e9f8bb362e418b0ed02f2a0bea5a9f6d1c739d